CLINICAL TRIAL: NCT03326063
Title: Therapeutic Control of Aspirin-Exacerbated Respiratory Disease
Brief Title: Therapeutic Control of Aspirin-Exacerbated Respiratory Disease With Ifetroban
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elliot Israel, MD, Director of Asthma Research Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017P001523
Record Dates: First submitted 2017-08-16; First posted 2017-10-30 (Actual); Results first posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: Nasal Polyps; Asthma, Aspirin-Induced; Aspirin-exacerbated Respiratory Disease; Aspirin-Sensitive Asthma With Nasal Polyps
MeSH Terms: conditions — Nasal Polyps; Asthma, Aspirin-Induced | interventions — ifetroban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ifetroban (Active Comparator): Subjects will be randomized to receive ifetroban (200 mg dose per day) for 4 weeks.
  Interventions: Drug: Ifetroban
- Placebo (Placebo Comparator): Subjects will be randomized to receive placebo for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ifetroban — 4-week, double-blind, placebo-controlled parallel-design trial of oral ifetroban (a TP receptor antagonist) in patients with AERD
  Other Names: ifetroban sodium
  Arms: Ifetroban
Drug: Placebo — 4-week, double-blind, placebo-controlled parallel-design trial of oral ifetroban (a TP receptor antagonist) in patients with AERD
  Arms: Placebo

SUMMARY:
The overall aim of the study is to determine the efficacy of oral ifetroban, a novel antagonist of T prostanoid (TP) receptors, as a treatment for patients with aspirin-exacerbated respiratory disease (AERD).

DETAILED DESCRIPTION:
The protocol involves a 4-week, double-blind, placebo-controlled parallel-design trial of oral ifetroban in patients with AERD. At the end of the 4-week treatment phase (ifetroban or placebo) each subject will undergo a graded oral aspirin desensitization procedure in order to initiate high-dose aspirin therapy, which is standard-of-care at our institution and is the only available therapy known to modify the course of AERD.

ELIGIBILITY:
Inclusion Criteria:

1. History of AERD, defined as meeting the diagnostic triad with:

   * History of physician-diagnosed asthma and
   * History of physician-diagnosed nasal polyposis and
   * History of pathognomonic reactions aspirin or other nonselective cyclooxygenase (COX) inhibitors.
2. Stable asthma (post-bronchodilator forced expiratory volume at one second (FEV1) of ≥70%, no glucocorticoid burst for at least 2 weeks prior to Visit 1, and no hospitalizations or ER visits for asthma for at least the prior 6 months)
3. Age between 18 and 70 years
4. No current smoking (not more than one instance of smoking in the last 3 months)
5. Non-pregnant

Exclusion Criteria:

1. Hypersensitivity to montelukast
2. Current use of zileuton
3. History of bleeding diathesis or use of anticoagulant or antiplatelet drugs
4. Current use of any NSAIDs aside from the aspirin provided during the study
5. Current use of beta blockers
6. Use of any biologics within the last 4 months prior to initiating the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Asthma Research Center, Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 38 potential participants were screened at Brigham and Women's Hospital.
Pre-assignment Details: 36 of whom underwent randomization per protocol, and 35 of whom completed the trial and were analyzed.
Groups:
- Ifetroban: Subjects will be randomized to receive ifetroban (200 mg dose per day) for 4 weeks.
  Ifetroban: 4-week, double-blind, placebo-controlled parallel-design trial of oral ifetroban (a thromboxane-prostanoid (TP) receptor antagonist) in patients with aspirin-exacerbated respiratory disease (AERD)
  Patients were then challenged to aspirin at ascending doses, starting at 40.5mg, 81mg, 162mg, and 325mg, given every 90 minutes until a reaction was provoked.
- Placebo: Subjects will be randomized to receive placebo for 4 weeks.
  Placebo: 4-week, double-blind, placebo-controlled parallel-design trial of oral ifetroban (a thromboxane-prostanoid (TP) receptor antagonist) in patients with aspirin-exacerbated respiratory disease (AERD)
  Patients were then challenged to aspirin at ascending doses, starting at 40.5mg, 81mg, 162mg, and 325mg, given every 90 minutes until a reaction was provoked.
Period: Overall Study
Arm/Group | Ifetroban | Placebo
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — COVID pandemic: subject recalled to her country | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ifetroban | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 16 | 16 | 32
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36
Provocative Dose 2 (PD2) During Aspirin Challenge [Mean (Standard Deviation); unit: mg] — Population: 36 subjects were randomized, but 1 subject in ifetroban arm was lost to follow-up and did not complete primary outcome for analysis.
  mg
    number analyzed (Participants) | 17 | 18 | 35
    (all) | 121 (48) | 142 (46) | 132 (47)

OUTCOME MEASURES:

1. Primary Outcome: Provocative Dose 2 (PD2) During Aspirin Challenge
Description: The calculated dose of aspirin that induces an increase in the Total Nasal Symptom Score (TNSS) of 2 from the pre-aspirin challenge value, "PD2"
  TNSS: A higher TNSS score suggests more severe symptoms, on a scale from 0-65 PD2: A higher PD2 suggests that the patient's threshold of reactivity of aspirin was higher
Time Frame: 6 weeks from screening visit ( at visit 2)
Measure: Mean (Standard Error); unit: mg
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 17 | 18
mg | 121 (48) | 142 (46)

2. Secondary Outcome: Percentage Change From Baseline of FEV1 During Aspirin Challenge (Bronchoconstriction)
Description: Severity of bronchoconstriction during the aspirin-induced reaction at Visit 2, compared between patients on placebo vs ifetroban, with the changes also analyzed with provocative aspirin dose as a covariate. Measured by an aspirin-induced decrease in FEV1.
Time Frame: At Visit 2. The change in FEV1 from the morning baseline to the aspirin-induced lowest value in FEV1 during reaction to aspirin challenge later that same day.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Ifetroban: Subjects randomized to receive Ifetroban.
- Placebo: Subjects randomized to receive placebo.
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 17 | 18
percentage change from baseline | -18.8 (3.6) | -8.4 (2.1)

3. Secondary Outcome: Aspirin-induced Leukotriene E4 (LTE4) Levels
Description: Increase of urinary levels of LTE4 during aspirin-induced reaction from Visit 2 pre-aspirin levels, compared between patients on placebo vs ifetroban, with the changes also analyzed with provocative aspirin dose as a covariate. LTE4 levels were calculated in a specialized laboratory.
Time Frame: Visit 2. The change in LTE4 levels from the morning baseline to the aspirin-induced highest value in LTE4 during reaction to aspirin challenge that same day.
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 17 | 18
ng/mg creatinine | 0.72 (0.30) | 0.15 (0.10)

4. Secondary Outcome: Change in Chronic Disease Control by Measurement of Lung Function Through FEV1
Description: Change from Visit 1 in baseline FEV1,compared between patients on placebo vs ifetroban.
Time Frame: 1 month (between Visit 1 and Visit 2)
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 17 | 18
percent change from baseline | -0.2 (1.3) | -0.5 (1.2)

5. Secondary Outcome: Change in Chronic Disease by Measurement of Asthma Control Through Asthma Control Questionnaire (ACQ) Score
Description: Change from Visit 1 in baseline ACQ (Asthma Control Questionnaire) score, compared between patients on placebo vs ifetroban.
  ACQ is a patient-reported questionnaire measurement of asthma control from 0-6, where lower scores suggest better asthma control. The score is the average result of the answer choices picked by the patient.
Time Frame: 1 month (between Visit 1 and Visit 2)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 17 | 18
scores on a scale | 0.17 (0.16) | -0.03 (0.11)

6. Secondary Outcome: Clinical Improvement of Chronic Disease - Sino-Nasal Outcome Test (SNOT-22) Score
Description: Change from Visit 1 in baseline SNOT-22 score at Visit 2, compared between patients on placebo vs ifetroban.
  The SNOT-22 is a patient-reported questionnaire with a summed scale that goes from 0-110 and a lower score suggests better sinonasal control.
Time Frame: 1 month (between Visit 1 and Visit 2)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 17 | 18
scores on a scale | 1.5 (3.0) | -2.0 (2.3)

7. Secondary Outcome: Fractional Exhaled Nitric Oxide (FeNO)
Description: Change from Visit 1 in baseline FeNO levels at Visit 2, compared between patients on placebo vs ifetroban.
Time Frame: 1 month (between Visit 1 and Visit 2)
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 17 | 18
parts per billion | 7.9 (9.0) | -3.4 (3.0)

8. Other Pre Specified Outcome: Percent Change in Urinary Eicosanoid (TXB2 and LTE4) Levels
Description: Change in levels of other urinary eicosanoids,from Visit 1 to Visit 2 pre-aspirin challenge and Visit 2 pre-aspirin to during the aspirin-induced reaction at Visit 2, compared between patients on placebo vs ifetroban, with the changes also analyzed with provocative aspirin dose as a covariate. Measurements include urinary thromboxane B2 (TXB2) and LTE4.
Time Frame: 1 month (between Visit 1 and Visit 2) and 6 weeks from screening visit ( at visit 2)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Nasal Eicosanoid Changes
Description: Change in levels of nasal eicosanoids, from Visit 1 to Visit 2 pre-aspirin challenge and Visit 2 pre-aspirin to during the aspirin-induced reaction at Visit 2, compared between patients on placebo vs ifetroban, with the changes also analyzed with provocative aspirin dose as a covariate.
Time Frame: 1 month (between Visit 1 and Visit 2) and 6 weeks from screening visit ( at visit 2)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Plasma/Serum Tryptase Changes
Description: Change in levels of plasma/serum tryptase, from Visit 1 to Visit 2 pre-aspirin challenge and Visit 2 pre-aspirin to during the aspirin-induced reaction at Visit 2, compared between patients on placebo vs ifetroban, with the changes also analyzed with provocative aspirin dose as a covariate.
Time Frame: 1 month (between Visit 1 and Visit 2) and 6 weeks from screening visit ( at visit 2)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Nasal Tryptase Changes
Description: Change in levels of nasal tryptase, from Visit 1 to Visit 2 pre-aspirin challenge and Visit 2 pre-aspirin to during the aspirin-induced reaction at Visit 2, compared between patients on placebo vs ifetroban, with the changes also analyzed with provocative aspirin dose as a covariate.
Time Frame: 1 month (between Visit 1 and Visit 2) and 6 weeks from screening visit ( at visit 2)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Platelet Activation - Numbers of Activated Platelets
Description: Change in numbers of activated platelets in the peripheral blood from Visit 1 to Visit 2 baseline (pre-aspirin administration) and during the aspirin-induced reaction at Visit 2 from Visit 2 baseline, compared between patients on placebo vs ifetroban, with the changes also analyzed with provocative aspirin dose as a covariate.
Time Frame: 1 month (between Visit 1 and Visit 2) and during aspirin challenge visit
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Platelet Activation - Percentages of Activated Platelets
Description: Change in percentages of activated platelets in the peripheral blood from Visit 1 to Visit 2 baseline (pre-aspirin administration) and during the aspirin-induced reaction at Visit 2 from Visit 2 baseline, compared between patients on placebo vs ifetroban, with the changes also analyzed with provocative aspirin dose as a covariate.
Time Frame: 1 month (between Visit 1 and Visit 2) and 6 weeks from screening visit ( at visit 2)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Platelet Activation - Numbers of Platelet-leukocyte Aggregates
Description: Change in numbers of platelet-leukocyte aggregates in the peripheral blood from Visit 1 to Visit 2 baseline (pre-aspirin administration) and during the aspirin-induced reaction at Visit 2 from Visit 2 baseline, compared between patients on placebo vs ifetroban, with the changes also analyzed with provocative aspirin dose as a covariate.
Time Frame: 1 month (between Visit 1 and Visit 2) and 6 weeks from screening visit ( at visit 2)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Platelet Activation - Percentages of Platelet-leukocyte Aggregates
Description: Change in percentages of platelet-leukocyte aggregates in the peripheral blood from Visit 1 to Visit 2 baseline (pre-aspirin administration) and during the aspirin-induced reaction at Visit 2 from Visit 2 baseline, compared between patients on placebo vs ifetroban, with the changes also analyzed with provocative aspirin dose as a covariate.
Time Frame: 1 month (between Visit 1 and Visit 2) and 6 weeks from screening visit ( at visit 2)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of randomized subject enrollment through study completion, about 8 weeks.
Groups:
- Placebo: Subjects with AERD who received Placebo
- Ifetroban: Subjects with AERD who received Ifetroban
Arm/Group | Placebo | Ifetroban
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 11/18 | 12/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Ifetroban (N=18)
Upper Respiratory Tract Infection/Sinusitis, Grade 2 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pregnant partner (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Rash, maculo-papular, Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Ear Pain, Grade 1 (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Stomach Pain, Grade 1 (Gastrointestinal disorders) | 1 (1) | 0 (0) — Includes vomiting, diarrhea, and/or constipation
Eye disorder- Stye, Grade 1 (Eye disorders) | 0 (0) | 1 (1)
Systemic reaction to aspirin challenge with extrapulmonary symptoms (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Lung Infection (influenza B-related pneumonia), Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
Wheezing, Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus disorder (bloody nose), Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bruising, Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Otitis Media, Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
Constipation, Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasal Congestion, Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage, Grade 1 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting, Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT03326063/Prot_SAP_000.pdf